CLINICAL TRIAL: NCT00004100
Title: Gemcitabine and Vinorelbine vs Standard Chemotherapy Containing Cisplatin for Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: Chemotherapy in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istituto Nazionale per lo Studio e la Cura dei Tumori (Other)
Collaborators: NCIC Clinical Trials Group (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067316; ITA-GEMVIN; CAN-NCIC-BR14; EU-99016
Record Dates: First submitted 1999-12-10; First posted 2004-04-16 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2008-06

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Gemcitabine; Vinorelbine

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which regimen of chemotherapy is more effective for non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two regimens of chemotherapy in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare gemcitabine plus vinorelbine vs standard chemotherapy containing cisplatin in terms of the effect on the quality of life of patients with stage IIIB or IV non-small cell lung cancer. II. Compare the effect of these regimens on the overall survival of these patients. III. Compare the toxic effects of these regimens in these patients. IV. Compare the effect of these regimens on the rate of objective response in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, stage of disease (IIIB vs IV), and performance status (0 vs 1 vs 2). Patients are randomized to one of two treatment arms. Arm I: Patients receive cisplatin IV on day 1 and either gemcitabine IV or vinorelbine IV on days 1 and 8. Arm II: Patients receive gemcitabine IV and vinorelbine IV on days 1 and 8. Treatment repeats every 21 days for up to 6 courses. Quality of life is assessed prior to therapy and before each course of chemotherapy to the fourth course.

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven non-small cell lung cancer Stage IV OR Stage IIIB with supraclavicular lymph node metastases and/or pleural effusion that is not curable with radiotherapy Measurable or evaluable disease No CNS metastases

PATIENT CHARACTERISTICS: Age: Under 70 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Neutrophil count at least 2000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: (Unless caused by liver metastases) Bilirubin no greater than 1.25 times upper limit of normal (ULN) SGOT or SGPT no greater than 1.25 times ULN Renal: Creatinine no greater than 1.25 times ULN Other: No prior or concurrent malignancy except basal or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Concurrent palliative radiotherapy allowed Surgery: Not specified

Max Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-11

CONTACTS AND LOCATIONS:
Overall Officials: Cesare Gridelli, MD, Study Chair — Istituto Nazionale per lo Studio e la Cura dei Tumori; Vera Hirsh, MD, FRCPC, Study Chair — Royal Victoria Hospital - Montreal
Locations (29):
- Italy (29):
  - Ospedale San Lazzaro, Alba
  - Ospedale Civile Avellino, Avellino
  - Ospedale G. Di Maria - Avola (SR), Avola (SR)
  - Azienda Ospedaliena G. Rummo, Benevento
  - Ospedale Cardarelli - Campobasso, Campobasso
  - Ospedale Civile Cosenza, Cosenza
  - Ospedale San Martino/Cliniche Universitarie Convenzionate, Genoa
  - Ospedale Gen. Provinciale Santa Maria Goretti, Latina
  - Ospedale di Legnano, Legnano
  - Ospedale Maggiore Lodi, Lodi
  - Ospedale Di Gabargnate Milanese, Milan
  - Ospedale San Carlo Borromeo, Milan
  - Istituto Di Science Biomediche San Paolo, Milan
  - Federico II University Medical School, Naples
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Ospedale S. Gennora USL 42, Naples
  - Ospedale Vincenzo Monaldi, Napoli
  - ASL 2 - Napoli, Napoli
  - Universita di Palermo, Palermo
  - Ospedale La Maddalena - Palermo, Palermo
  - Ospedale S. Francesco - Paola, Paola (CS)
  - Ospedale Agnelli, Pinerolo
  - Ospedale San Carlo, Potenza
  - Ospedali Riuniti, Reggio Calabria
  - U.S.S.L. 33, Rho
  - Ospedale Oncologieo G. Fortunato, Rionero Sannitico
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
  - Ospedale Civile - Rovereto, Rovereto
  - Ospedale San Bortolo, Vicenza

REFERENCES:
- [Background] Wheatley-Price P, Le Maître A, Ding K, et al.: The influence of sex on efficacy, toxicity and delivery of treatment in National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) non-small cell lung cancer (NSCLC) chemotherapy trials. [Abstract] J Clin Oncol 26 (Suppl 15): A-8054, 2008.
- [Result] Gridelli C, Gallo C, Shepherd FA, Illiano A, Piantedosi F, Robbiati SF, Manzione L, Barbera S, Frontini L, Veltri E, Findlay B, Cigolari S, Myers R, Ianniello GP, Gebbia V, Gasparini G, Fava S, Hirsh V, Bezjak A, Seymour L, Perrone F. Gemcitabine plus vinorelbine compared with cisplatin plus vinorelbine or cisplatin plus gemcitabine for advanced non-small-cell lung cancer: a phase III trial of the Italian GEMVIN Investigators and the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2003 Aug 15;21(16):3025-34. doi: 10.1200/JCO.2003.06.099. Epub 2003 Jul 1. PMID 12837810
- [Result] Gridelli C, Shepherd F, Perrone F, et al.: Gemvin III: a phase III study of gemcitabine plus vinorelbine (GV) compared to cisplatin plus vinorelbine or gemcitabine chemotherapy (PCT) for stage IIIb or IV non-small cell lung cancer (NSCLC): an Italo-Canadian study. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1165, 2002.